CLINICAL TRIAL: NCT00836069
Title: A Phase 3, Randomized, Double-Blind, Parallel Group, 10-Week Placebo Controlled Fixed Dose Study of PD 0332334 and Paroxetine Evaluating the Efficacy and Safety of PD 0332334 for the Treatment of Generalized Anxiety Disorder
Brief Title: Fixed Dose Study of PD 0332334 and Paroxetine for the Treatment of Generalized Anxiety Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pfizer has terminated the execution of this protocol
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Itai Danovitch, Chair, Department of Psychiatry and Behavioral Neurosciences, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15002
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Disorders
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PD 0332334-α2δ ligand (450mg) (Experimental): PD 0332334, 450mg/day, for 8 weeks and then 2 weeks of dose tapering.
  Interventions: Drug: No drug name provided by Sponsor; drug referenced as PD 0332334
- PD 0332334-α2δ ligand (600mg) (Experimental): PD 0332334, 600mg/day, for 8 weeks and then 2 weeks of dose tapering.
  Interventions: Drug: No drug name provided by Sponsor; drug referenced as PD 0332334
- Paroxetine (Active Comparator): Paroxetine, 20mg/daym for 8 weeks and then 2 weeks of dose tapering.
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): Inactive Substance (placebo) for 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: No drug name provided by Sponsor; drug referenced as PD 0332334 — Experimental study drug for generalized anxiety disorder, oral tablet, at a total daily dose of 450mg or 600mg, twice daily for 8 weeks and then 2 weeks of dose tapering.
  Arms: PD 0332334-α2δ ligand (450mg); PD 0332334-α2δ ligand (600mg)
Drug: Paroxetine — FDA Approved medication for generalized anxiety disorder, oral tablet, at 20mg, once daily for 8 weeks and then 2 weeks of dose tapering.
  Other Names: Paxil, Paxil CR, Brisdelle, and Pexeva
  Arms: Paroxetine
Drug: Placebo — inactive substance, oral tablet, once per day, for 10 weeks.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, parallel-group, multi-site, Phase 3, placebo controlled fixed-dose study of PD 0332334 and paroxetine in 528 outpatients with generalized anxiety disorder. Subjects will be randomized to the following treatments (132 subjects per treatment group):

PD 0332334 225 mg twice a day (450 mg/day), PD 0332334 300 mg twice a day (600 mg/day), placebo once a day in the morning or paroxetine 20 mg once a day in the morning (20 mg/day).

DETAILED DESCRIPTION:
The study will consist of 3 phases: an initial screening phase which must be completed 7 to 14 days prior to randomization; an 8-week double-blind treatment phase; and a 2-week double-blind dose-tapering follow-up phase. After obtaining written informed consent the investigator will initiate washout of prior psychotropic medications. After the washout of prior psychotropic medications has been completed the investigator must ensure that the subject is no longer taking psychotropic medication for at least 14 days prior to the randomization visit. In addition the investigator must ensure that screening visit procedures (with the exception of obtaining informed consent) are completed within 14 days of the randomization visit.

Potential subjects will be approached during a regularly scheduled clinic visit, upon referral from another physician, or in response to research advertisements. Those who call in will participate in a short phone pre-screen. This allows us to determine if the person fits the most limiting inclusion/exclusion criteria before requesting they dedicate a longer period of time for an in-person screen. Additionally it gives interested individuals the opportunity to learn more about the study and to review the consent form with family, friends, and other physicians prior to coming in for the screen and making a final decision regarding study enrollment. Once the subject has given informed consent, the screening process for the study will commence.

Subjects who fulfill entry criteria will be randomized to receive ONE of the following 4 treatments in a double-blind fashion: PD 0332334 225 mg twice a day, PD 0332334 300 mg twice a day, placebo, and paroxetine 20 mg once in the morning. PD 0332334 will be titrated up in the PD 0332334 225 mg twice a day and PD 0332334 300 mg twice daily treatment groups. The titration of PD 0332334 will be from 125 mg in the beginning of the study. In addition the PD 0332334 225 mg twice a day and PD 0332334 300 mg twice a day treatment groups will be titrated down at the end of the study. The 20 mg daily dose of paroxetine used in this study is based on the approved label for the use of paroxetine in patients with generalized anxiety disorder. Doses were selected for this Phase 3 study based on safety and efficacy information known about PD 0332334 and pregabalin, an α2δ ligand approved for the treatment of generalized anxiety disorder in Europe

The subjects enrolled will be men and women ages 18 to 65 who meet DSM-IV criteria for generalized anxiety disorder with a preponderance of anxious symptoms over depressive symptoms.

De-identified blood samples will be collected from study subjects at Screening (Visit 1) according to the standard Molecular Profiling supplement to the protocol. Participation in this component is optional for study subjects. Samples may be utilized in the future to investigate generalized anxiety disorder genetics, expression metabonomics and protein biomarker profiles, drug-response, or other genetic or biomarker questions. [Metabonomics: The study of metabolic responses to drugs, environmental changes and diseases. Metabonomics is an extension of genomics (concerned with DNA) and proteomics (concerned with proteins). ]

Additionally, partners of male participants who become pregnant during the course of the study, will be requested to participate in order for the sponsor to collect safety information and understand the effects, if any, that PD 0332334 may have on her pregnancy or the fetus. Details of the this sub-study are described in the separate 'pregnant partner' consent form. Pregnant partners will be be asked to sign a separate HIPAA and consent form in order to participate.

The investigators have recently received notification of an serious adverse event at another site that has already begun recruitment for this study. The MediWatch report for that serious adverse event is included as a Supporting document on WEBRIDGE. Additionally, a protocol change clarifying the procedures to collect lab information to calculate the estimate Creatinine Clearance has been submitted. This document has been added as a supporting document on WEBRIDGE (IRB web-based management portal).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Diagnosis of generalized anxiety disorder (Diagnostic and Statistical Manual-IV [DSM-IV], 300.02) as established by the clinician.
2. Subjects must have a Hamilton-A total score ≥20 at the screening (V1) and randomization (V2) visits. Subjects must also have a Covi Anxiety Scale score of ≥9 and a Raskin Depression Scale score ≤7 at the Screening (V1) visit to ensure predominance of anxiety symptoms over depression symptoms.
3. Otherwise healthy men or non-pregnant, non-lactating women (women must be using a hormonal or barrier method of contraception or be postmenopausal or surgically sterilized). Healthy is defined as no other clinically relevant abnormalities identified by a detailed medical history, full physical examination including sitting blood pressure and heart rate measurement, 12-lead ECG, and clinical laboratory tests.
4. Age 18 to 65 years, inclusive.
5. All women must have negative pregnancy tests at the Screening (Visit 1) and Randomization (Visit 2) visits.
6. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
7. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, neurologic, active infections, immunological, or allergic disease (including drug allergies).
2. Any of the following current (within the past 6 months through the present) Diagnostic and Statistical Manual of Mental Disorders-IV Axis I diagnoses:

   * Major depressive disorder;
   * Obsessive compulsive disorder;
   * Panic disorder;
   * Agoraphobia;
   * Posttraumatic stress disorder;
   * Anorexia;
   * Bulimia;
   * Caffeine-induced anxiety disorder;
   * Alcohol or substance abuse or dependence unless in full remission for at least 6 months;
   * Social anxiety disorder.
3. Any of the following past or current Diagnostic and Statistical Manual of Mental Disorders-IV Axis I diagnoses:

   * Schizophrenia;
   * Psychotic disorder;
   * Delirium, dementia, amnestic, and other clinically significant cognitive disorders;
   * Bipolar or schizoaffective disorder;
   * Cyclothymic disorder;
   * Dissociative disorders.
4. Antisocial or borderline personality disorder.
5. Serious suicidal risk per the clinical investigator's judgment. (Note: The Suicidality module of the Mini-Mental State Examination diagnostic interview and the Columbia-Suicide Severity Rating Scale should be used as aids to the assessment of suicidality, but do not replace overall clinical judgment in determination of suicidal risk).
6. Current use of psychotropic medications (ie, drugs normally prescribed for depression, mania, anxiety, insomnia, or psychosis) that cannot be discontinued 2 weeks prior to randomization. Fluoxetine is prohibited within 5 weeks of randomization. In the event of inadvertent administration of psychotropic medications during the 2 weeks prior to randomization, continued eligibility will be assessed on a case by case basis by the investigator and the medical monitor.
7. Use of drugs, supplements, prescription or nonprescription, or food that have psychoactive properties. In the event of inadvertent use of such products during the 2 weeks prior to randomization, continued eligibility will be assessed on a case by case basis by the investigator and the medical monitor. In addition, following a discussion of the individual case between the medical monitor and the investigator, the medical monitor may allow minimal anxiolytic medication (for example a benzodiazepine) use for subjects who experience significant intolerable anxiety during the final week of the study (Days 64-71).
8. Subjects who have been treated with monoamine oxidase inhibitors in the 14 days prior to the baseline visit.
9. Regular use of benzodiazepines during the 3 months prior to Screening (for at least 5 out of 7 days per week).
10. Subjects initiating formal psychotherapy within 3 month prior to screening who intend to continue formal psychotherapy during the study. This includes psychodynamic, cognitive, and interpersonal therapies.
11. Positive drug tests at Screening (Visit 1) or Randomization (Visit 2) visits for any of the following substances or classes of compounds: amphetamines, barbiturates, opiates, benzodiazepines, sedatives and hypnotics, cocaine, phencyclidine (PCP), cannabinoids, or other illegal or illicit drugs. An exception to the exclusion for a positive benzodiazepine, opiate, or sedative and hypnotic drug test at the Screening (Visit 1) visit may be granted by the Pfizer medical monitor if written evidence of a valid, current prescription is presented.
12. Any condition possibly affecting drug absorption (eg, gastrectomy).
13. Subjects with a current seizure disorder.
14. Subjects with a history of life-threatening neoplasms within 5 years prior to study entry, other than carcinoma in situ of the cervix or basal cell carcinoma of the skin.
15. Subjects with hypothyroidism or hyperthyroidism, except subjects who are euthyroid and have been on stable doses of thyroid replacement for 6 months or more.
16. Subjects with any clinically unstable hematological, autoimmune, endocrine, neurological, renal, hepatic, retinal, gastrointestinal, or cardiovascular disorder.
17. Subjects with uncontrolled narrow angle glaucoma.
18. Subjects with a known hypersensitivity to paroxetine.
19. History of allergy or intolerance to paroxetine.
20. Subjects with a prior history of insufficient response to paroxetine in the treatment of generalized anxiety disorder (with an adequate trial of therapy).
21. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception for the duration of the study.
22. Treatment with an investigational drug within 60 days preceding the first dose of trial medication.
23. Estimated creatinine clearance <55 mL/min (using Cockcroft-Gault equation).
24. Alanine aminotransferase or aspartate aminotransferase (AST) levels >3 times the upper limit of normal at Screening (Visit 1).
25. Male and Female subjects with a screening 12-lead ECG demonstrating QTcF (Fredericia's correction) >450 msec, if confirmed with an unscheduled repeat 12-lead ECG's at the screen visit. In the event of discrepant QTcF values (i.e., >450 msec and <450 msec) after repeat unscheduled 12-lead ECG at screen, a decision with regards protocol eligibility will be made on a case by case basis between the investigator and medical monitor.
26. History of lack of efficacy for treatment of generalized anxiety disorder with, or allergy or intolerance to, other α2δ drugs (pregabalin, gabapentin).
27. Blood donation of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
28. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | Every Week for 10 weeks
  The purpose of administering the scale is to analyze the severity of the patient's anxiety and will take approximately 10 to 15 minutes to administer.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center Department of Psychiatry and Behavioral Neurosciences, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No